CLINICAL TRIAL: NCT01179438
Title: Effect of Dexmedetomidine on Microcirculation in Patients Undergoing Extracorporeal Shock Wave Lithotripsy
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Yu-Chang Yeh, National Taiwan University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 201003036M
Record Dates: First submitted 2010-08-09; First posted 2010-08-11 (Estimated); Last update posted 2012-12-10 (Estimated); Status verified 2010-06

CONDITIONS: Microcirculation
MeSH Terms: interventions — Dexmedetomidine

INTERVENTIONS:
Drug: Dexmedetomidine — The loading does of 0.5 mcg/kg dexmedetomidine is infused over 10 minutes. The following maintenance does of dexmedetomidine is 0.5 mcg/kg/hour.

SUMMARY:
Dexmedetomidine administration for minor procedure, such as extracorporeal shock wave lithotripsy, provides good quality of sedation and analgesia. Dexmedetomidine is a highly selective α2-adrenergic receptor agonist which causes sedative effects and reduces opioid requirements in the perioperative period. Extracorporeal shock wave lithotripsy may cause pain and result in tachycardia and vasoconstriction-related hypertension. Surgical or procedural stress may induce inflammation and it may cause further microthrombosis. Both vasoconstriction and microthrombosis will alter the microcirculatory status. Dysfunction of microcirculation may impair tissue perfusion and result in organ dysfunction. Dexmedetomidine may induce vasodilation by slow intravenous infusion for sedation. Dexmedetomidine may also reduce inflammation. After reviewing the literature, the investigators found that the effect of dexmedetomidine on microcirculation was not well investigated. By application of the non-invasive technique of sidestream dark field imaging, the investigators can investigate the vessel density, percentage of perfused vessels, and microvascular flow index on sublingual vessels.

The goal of this study is to identify the effect of dexmedetomidine on sublingual microcirculation in patient undergoing extracorporeal shock wave lithotripsy.

ELIGIBILITY:
Inclusion Criteria:

* Patient who is older than 18 years old and less than 75 years old
* Patient who receive extraproporeal shock wave lithotripsy with ASA class I or II
* Patient who has understood the inform consent and agree to participate this study

Exclusion Criteria:

* Patient's hemodynamic status is unstable in spite of adequate management or presence of signs of shock
* Patient who has a past history of allergy to s dexmedetomidine
* Patient who has history of cardiovascular, renal or hepatic dysfunction
* Patient who has participated in any other investigational study of other drugs currently
* Female patient who is pregnant or considers breast feeding currently
* Patient who has suspected full stomach

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2011-06 (Estimated); Study Completion 2011-06 (Estimated)

PRIMARY OUTCOMES:
Microcirculation status | 120min
  Microcirculation examination

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, anesthesiology department, Taipei, Taiwan